CLINICAL TRIAL: NCT03464045
Title: Post-authorisation Safety Study to Assess the Risk of Urinary Tract Malignancies in Relation to Empagliflozin Exposure in Patients With Type 2 Diabetes: a Multi-database European Study
Brief Title: Empa PASS on Urinary Tract Malignancies
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0097
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Empagliflozin initiators - UK: Participants with Type 2 diabetes mellitus (T2D) initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2021 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from Clinical Practice Research Datalink (CPRD) (General practitioner Online Data [GOLD], and Aurum) in the United Kingdom (UK).
  Interventions: Drug: empagliflozin
- DPP4-i initiators - UK: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2021 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from CPRD (General practitioner Online Data [GOLD], and Aurum) in the UK.
  Interventions: Drug: DPP-4 inhibitors
- Empagliflozin initiators - Sweden: Participants with T2D initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Sweden.
  Interventions: Drug: empagliflozin
- DPP4-i initiators - Sweden: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Sweden.
  Interventions: Drug: DPP-4 inhibitors
- Empagliflozin initiators - Finland: Participants with T2D initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Finland.
  Interventions: Drug: empagliflozin
- DPP4-i initiators - Finland: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Finland.
  Interventions: Drug: DPP-4 inhibitors

INTERVENTIONS:
Drug: empagliflozin — empagliflozin
  Groups: Empagliflozin initiators - Finland; Empagliflozin initiators - Sweden; Empagliflozin initiators - UK
Drug: DPP-4 inhibitors — DPP-4 inhibitors
  Groups: DPP4-i initiators - Finland; DPP4-i initiators - Sweden; DPP4-i initiators - UK

SUMMARY:
The aim of the study is to assess the risk of urinary tract malignancies in patients initiating empagliflozin (free or fixed dose combination) compared to patients initiating a dipeptidyl peptidase-4 (DPP-4) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Age over 18 years at index date
* At least 1 year of membership in the medication database prior to index date

Exclusion Criteria:

* Patients with any cancer (excluding non-melanoma skin cancer) recorded at any time prior to the index date (i.e. during the available look-back time)
* Diagnosis of type 1 diabetes or other specific non-type 2 diabetes
* Use of any SGLT-2 inhibitor or any DPP-4 inhibitor (including free and fixed-dose combinations) recorded at any time prior to index date (i.e. during the available look-back time).
* Use of fixed-dose combinations of SGLT-2 inhibitors with DPP-4 inhibitors
* Diagnosis of end stage renal disease or receipt of renal dialysis recorded at any time prior to index date (i.e. during the available look-back time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational, comparative, cohort safety study based on European healthcare databases and includes databases from the UK, Finland, and Sweden.
Sampling Method: Probability Sample
Enrollment: 344995 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Korhonen, 358-50-3652990, Principal Investigator — pasi.korhonen@epidresearch.com
Locations (3):
- The National Register Data, Helsinki, Finland
- The Swedish prescribed drug register, Stockholm, Sweden
- United Kingdom Clinical Practice Research Datalink (CPRD), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, comparative, cohort-based Post-authorisation-safety study (PASS) to assess the risk of urinary tract malignancies in patients affected by type 2 diabetes mellitus initiating empagliflozin or dipeptidyl peptidase-4 inhibitor (DPP-4i) between 1-Aug-2014 and 31-Dec-2021 in the United Kingdom (UK), Sweden, and Finland.
Pre-assignment Details: Throughout the study, different data extraction timepoints were used, starting from 2016 to 2023, and retrospective data was analyzed. Only subjects that met all inclusion and none of the exclusion criteria were included.
Period: Overall Study
Arm/Group | Empagliflozin Initiators - UK | DPP4-i Initiators - UK | Empagliflozin Initiators - Sweden | DPP4-i Initiators - Sweden | Empagliflozin Initiators - Finland | DPP4-i Initiators - Finland
Started | 27410 | 123334 | 35954 | 73623 | 21942 | 62732
Completed | 27410 | 123334 | 35954 | 73623 | 21942 | 62732
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population: population before propensity score-matching.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin Initiators - UK | DPP4-i Initiators - UK | Empagliflozin Initiators - Sweden | DPP4-i Initiators - Sweden | Empagliflozin Initiators - Finland | DPP4-i Initiators - Finland | Total
Number analyzed (Participants) | 27410 | 123334 | 35954 | 73623 | 21942 | 62732 | 344995
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.51 (10.96) | 63.50 (13.24) | 62.75 (11.18) | 66.65 (12.66) | 60.11 (11.84) | 66.04 (13.42) | 63.78 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16922 | 72124 | 24825 | 44352 | 13048 | 34233 | 205504
  Male | 10488 | 51210 | 11129 | 29271 | 8894 | 28499 | 139491
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Urinary Tract Cancer
Description: Occurrence of urinary tract cancer, which include malignant neoplasm and carcinoma in situ of the urinary tract, is reported as incidence rates per 1000 patient years. Incidence rates were estimated using Poisson regression and computed as the number of outcome events divided by the total person-time-at-risk (in years), multiplied by 1,000 for easier comparison. The country-level datasets were analyzed separately. Thereafter, pooled incidence rates were estimated using the aggregated number of outcome events and time-at-risk of all study countries using the Poisson regression.
Time Frame: From 181 days after index date until the occurrence of a censoring event or cancer outcome event. Up to 6 (Sweden/Finland) or 7 years (UK).
Population: Main analysis population: participants that were matched using propensity scores (PS) conditional on variables such as index date, disease progression, comorbidities, treatment history, age, and sex; and who did not have observations of any censoring events or outcome cancer events within the latency period (spanning 180 days after the index date).
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient years
Groups:
- Empagliflozin Initiators - UK, PS-matched: Participants with Type 2 diabetes mellitus (T2D) initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2021 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from Clinical Practice Research Datalink (CPRD) (General practitioner Online Data [GOLD], and Aurum) in the United Kingdom (UK).
  The cohort was propensity scored-matched.
- DPP4-i Initiators - UK, PS-matched: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2021 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from CPRD (General practitioner Online Data [GOLD], and Aurum) in the UK.
  The cohort was propensity scored-matched.
- Empagliflozin Initiators - Sweden, PS-matched: Participants with T2D initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Sweden.
  The cohort was propensity scored-matched. As no patients initiated empagliflozin treatment in 2014 in Sweden, DPP-4i initiators in 2014 were excluded from PS matching.
- DPP4-i Initiators - Sweden, PS-matched: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Sweden.
  The cohort was propensity scored-matched. As no patients initiated empagliflozin treatment in 2014 in Sweden, DPP-4i initiators in 2014 were excluded from PS matching.
- Empagliflozin Initiators - Finland, PS-matched: Participants with T2D initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Finland.
  The cohort was propensity scored-matched. As no patients initiated empagliflozin treatment in 2014 in Finland, DPP-4i initiators in 2014 were excluded from PS matching.
- DPP4-i Initiators - Finland, PS-matched: Participants with T2D initiating (first purchase/prescription) a dipeptidyl peptidase-4 inhibitor (DPP-4i) (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the nationwide registers in Finland.
  The cohort was propensity scored-matched. As no patients initiated empagliflozin treatment in 2014 in Finland, DPP-4i initiators in 2014 were excluded from PS matching.
- Empagliflozin Initiators - All Countries, PS-matched: This arm includes all the empagliflozin initiators in the propensity scored-matched cohorts.
  Participants with T2D initiating (first purchase/prescription) empagliflozin (study drug), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2021 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the CPRD (General practitioner Online Data [GOLD], and Aurum) in the UK, and from the from the nationwide registers in Sweden and Finland. As no patients initiated empagliflozin treatment in 2014 in Sweden and Finland, DPP-4i initiators in 2014 were excluded from PS matching.
- DPP4-i Initiators - All Countries, PS-matched: This arm includes all the DPP4-i initiators in the propensity scored-matched cohorts.
  Participants with T2D initiating (first purchase/prescription) a DPP-4i (comparator), in free form or in fixed-dose combination with metformin, between 1-Aug-2014 and 31-Dec-2020 (index date), and with more than 6 months of possible follow-up (index date less than 6 months prior to end of study date). The study population was identified from the CPRD (General practitioner Online Data [GOLD], and Aurum) in the UK, and from the from the nationwide registers in Sweden and Finland. As no patients initiated empagliflozin treatment in 2014 in Sweden and Finland, DPP-4i initiators in 2014 were excluded from PS matching.
Arm/Group | Empagliflozin Initiators - UK, PS-matched | DPP4-i Initiators - UK, PS-matched | Empagliflozin Initiators - Sweden, PS-matched | DPP4-i Initiators - Sweden, PS-matched | Empagliflozin Initiators - Finland, PS-matched | DPP4-i Initiators - Finland, PS-matched | Empagliflozin Initiators - All Countries, PS-matched | DPP4-i Initiators - All Countries, PS-matched
Number analyzed (Participants) | 18838 | 44838 | 20844 | 25682 | 15696 | 25157 | 55378 | 95677
Events per 1000 patient years | 0.73 [0.46 to 1.16] | 1.07 [0.84 to 1.37] | 1.34 [0.95 to 1.89] | 1.52 [1.13 to 2.05] | 1.27 [0.86 to 1.87] | 1.49 [1.13 to 1.96] | 1.10 [0.88 to 1.38] | 1.29 [1.11 to 1.51]
Statistical Analysis 1: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; Crude HRs were calculated using a Cox proportional hazards model with as-treated exposure (continuous exposure to the study drugs, defined as having consecutive treatment episodes separated by a grace period of 30 days, starting from index date) as the only included variable. Country-level HRs were analyzed separately. Thereafter, random-effects meta-analyses were conducted to pool the HRs from all countries, accounting for potential heterogeneity between the country-level effect sizes; Test type: Other; p = 0.122, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.61 to 1.06] — Crude hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; Base HRs were calculated using a Cox proportional hazards model by adjusting for variables unbalanced after PS matching. To be included in the Cox model, each covariate is required to have a minimum of 5 events per category level to avoid converge failure. Country-level HRs were analyzed separately. Thereafter, random-effects meta-analyses were conducted to pool the HRs from all countries, accounting for potential heterogeneity between the country-level effect sizes; Test type: Other; p = 0.417, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.67 to 1.18] — Base hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; Adjusted HRs were calculated using a Cox proportional hazards model by adjusting for variables unbalanced after PS matching, and pre-specified time-varying covariates. To be included in the Cox model, each covariate is required to have a minimum of 5 events per category level. Country-level HRs were analyzed separately. Thereafter, random-effects meta-analyses were conducted to pool the HRs from all countries, accounting for potential heterogeneity between the country-level effect sizes; Test type: Other; p = 0.376, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.17] — Adjusted hazard ratio of empagliflozin/DPP-4i

2. Primary Outcome: Occurrence of Bladder Cancer
Description: Occurrence of bladder cancer, malignant and carcinoma in situ, is reported as incidence rates per 1000 patient years. Incidence rates were estimated using Poisson regression and computed as the number of outcome events divided by the total person-time-at-risk (in years), multiplied by 1,000 for easier comparison. The country-level datasets were analyzed separately. Thereafter, pooled incidence rates were estimated using the aggregated number of outcome events and time-at-risk of all study countries using the Poisson regression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient years
Arm/Group | Empagliflozin Initiators - UK, PS-matched | DPP4-i Initiators - UK, PS-matched | Empagliflozin Initiators - Sweden, PS-matched | DPP4-i Initiators - Sweden, PS-matched | Empagliflozin Initiators - Finland, PS-matched | DPP4-i Initiators - Finland, PS-matched | Empagliflozin Initiators - All Countries, PS-matched | DPP4-i Initiators - All Countries, PS-matched
Number analyzed (Participants) | 18838 | 44838 | 20844 | 25682 | 15696 | 25157 | 55378 | 95677
Events per 1000 patient years | 0.45 [0.25 to 0.81] | 0.67 [0.49 to 0.90] | 0.92 [0.61 to 1.40] | 1.03 [0.71 to 1.48] | 0.51 [0.27 to 0.94] | 0.64 [0.42 to 0.98] | 0.63 [0.47 to 0.85] | 0.74 [0.6 to 0.91]
Statistical Analysis 1: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.220, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.55 to 1.15] — Crude hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.628, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.63 to 1.32] — Base hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.632, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.63 to 1.33] — Adjusted hazard ratio of empagliflozin/DPP-4i

3. Primary Outcome: Occurrence of Renal Cancer
Description: Occurrence of malignant renal cancer is reported as incidence rates per 1000 patient years. Incidence rates were estimated using Poisson regression and computed as the number of outcome events divided by the total person-time-at-risk (in years), multiplied by 1,000 for easier comparison. The country-level datasets were analyzed separately. Thereafter, pooled incidence rates were estimated using the aggregated number of outcome events and time-at-risk of all study countries using the Poisson regression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient years
Arm/Group | Empagliflozin Initiators - UK, PS-matched | DPP4-i Initiators - UK, PS-matched | Empagliflozin Initiators - Sweden, PS-matched | DPP4-i Initiators - Sweden, PS-matched | Empagliflozin Initiators - Finland, PS-matched | DPP4-i Initiators - Finland, PS-matched | Empagliflozin Initiators - All Countries, PS-matched | DPP4-i Initiators - All Countries, PS-matched
Number analyzed (Participants) | 18838 | 44838 | 20844 | 25682 | 15696 | 25157 | 55378 | 95677
Events per 1000 patient years | 0.24 [0.11 to 0.54] | 0.34 [0.22 to 0.52] | 0.42 [0.22 to 0.78] | 0.50 [0.29 to 0.84] | 0.76 [0.46 to 1.26] | 0.82 [0.57 to 1.19] | 0.45 [0.32 to 0.65] | 0.51 [0.4 to 0.65]
Statistical Analysis 1: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.420, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.29] — Crude hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 2: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.606, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.57 to 1.38] — Base hazard ratio of empagliflozin/DPP-4i
Statistical Analysis 3: Comparison: Empagliflozin Initiators - UK, PS-matched vs DPP4-i Initiators - UK, PS-matched vs Empagliflozin Initiators - Sweden, PS-matched vs DPP4-i Initiators - Sweden, PS-matched vs Empagliflozin Initiators - Finland, PS-matched vs DPP4-i Initiators - Finland, PS-matched; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.609, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.57 to 1.38] — Adjusted hazard ratio of empagliflozin/DPP-4i

ADVERSE EVENTS:
Time Frame: This study used secondary data only. Hence, reporting of adverse reactions was not required nor possible.
Description: This study used secondary data only. Hence, reporting of adverse reactions was not required nor possible.
Arm/Group | Empagliflozin Initiators - UK | DPP4-i Initiators - UK | Empagliflozin Initiators - Sweden | DPP4-i Initiators - Sweden | Empagliflozin Initiators - Finland | DPP4-i Initiators - Finland
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03464045/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03464045/SAP_001.pdf